CLINICAL TRIAL: NCT03402620
Title: Starting Dose of Gonadotropin for Poor Responders in IVF Cycles
Brief Title: Poor Responders Infertile Patients -A Great Clinical Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- four ampoules group (Active Comparator): gonadotropin starting dose is 4 ampoules daily
  Interventions: Drug: Gonadotropins
- six ampoules group (Active Comparator): gonadotropin starting dose is 6 ampoules daily
  Interventions: Drug: Gonadotropins

INTERVENTIONS:
Drug: Gonadotropins — Human menopausal gonadotropin 75 IU ampoules start at cycle day 2

SUMMARY:
infertile , poor responders patients who underwent ICSI. The participants were divided into 2 groups according to the starting dose of Gn stimulation. Group I started with 4 ampoules while group II started with 6 ampoules

DETAILED DESCRIPTION:
Participants will be randomized to start induction with 4 or 6 ampoules of gonadotropins from day 2 till the day of human chorionic gonadotropin (HCG), dose adjusted according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by TVUS scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day 6 for folliculometry and endometrial thickness and pattern. Cetrotide (MerckSerono, Germany) 0.25 subcutaneously will be added when the leading follicle (DF) reaches >12 mm and HCG 10 000 IU intramuscularly (Pregnyl, Merck Sharp, United Kingdom)will be given only if we have at least 3 mature follicles >14 mm and the leading one >17 mm; then, ovum pickup (OPU) was done after 36 hours of HCG and metaphase II ocytes were analyzed. The intracytoplasmic sperm injection (ICSI) procedure will be performed in all cases to avoid low fertilization rate by conventional IVF. Fertilization was assessed 16 to 18 hours after ICSI, and embryo quality will be evaluated 2 and 3 days after ICSI according to the number of blastomeres and the degree of fragmentation and multinucleation. Oocytes were collected and embryos will be cultured in ISM1 culture medium (Origiomedicult media, Denmark). Transfer of cleaving embryos will be done on day 3 after oocyte retrieval (using Labotect semirigid catheter; labotect GmbH, Germany), when the woman has at least 1 embryo (GI) otherwise canceled embryo transfer (ET). The ET was done by 1 person in each center. Both of the transferring consultants have more than 5 years experience in IVF unit. . All patients will receive luteal support in the form of daily progesterone cyclogest (Actavis, United Kingdom) 800 mg daily starting from day of ovum retrieval till day of hCG testing. Serum b hCG level was assessed on day 14 after ET and considered positive if >5 mIU/ml. The TVUS was performed 28 days after ET to confirm ongoing pregnancy by visualization of intrauterine sac.

ELIGIBILITY:
Inclusion Criteria:

* Poor responders according to "Bologna consensus" with at least 2 of the following 3 points should be present:

  1. Age >40 years or other cause of poor function.
  2. AFC<2-5 in both ovaries or AMH < 0.5-1.1 ng/dl 2)
  3. History of poor response with conventional stimulation protocol

Exclusion Criteria:

1. Uterine factor.
2. Severe male factor.
3. Endometriosis.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
number of retrieved oocytes | 34 hours after HCG triggering
  The number of oocyte retrived at ovum pickup

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided